CLINICAL TRIAL: NCT04499547
Title: Effect of a YouTube-Delivered Physical Activity Intervention on College Students' Aerobic and Muscle-Strengthening Physical Activity: A Randomized Controlled Trial
Brief Title: YouTube-Delivered Physical Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2728
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: youtube; physical activity; fitness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity intervention (Experimental): Will receive twice-weekly, YouTube-delivered aerobic and muscle-strengthening physical activity videos for 8 weeks.
  Interventions: Behavioral: YouTube-delivered aerobic and muscle-strengthening physical activity intervention
- General health education control (No Intervention): Will receive twice-weekly, YouTube-delivered videos with general health education information for 8 weeks.

INTERVENTIONS:
Behavioral: YouTube-delivered aerobic and muscle-strengthening physical activity intervention — Participants in the intervention group will receive two YouTube-delivered videos each week, for 8 weeks. In detail, on Monday, participants will receive an aerobic-based physical activity video with information and a workout to complete and on Thursdays, the participants will receive a video with muscle-strengthening physical activity information and a workout to complete.
  Arms: Physical activity intervention

SUMMARY:
This study will be an 8-week randomized controlled trial examining the effects of a YouTube-delivered aerobic and muscle strengthening physical activity intervention on university students' physical activity, fitness, sleep quality, and psychosocial health outcomes. Participants will be randomized into 1 of 2 groups: (1) intervention group (receive twice-weekly YouTube videos [1 aerobic workout video; 1 muscle-strengthening workout video] for 8 weeks); or (2) control group (receive twice-weekly YouTube videos with general health information [no physical activity-related information or workouts] for 8 weeks). Baseline (0 weeks), mid-point (4 weeks), and post-test (8 weeks) testing will take place and the following outcome measures will be assessed at these time points: participants' free-living (7-day) objectively-measured physical activity and sleep quality data will be collected; anthropometric measures (height, weight, percent body fat); cardiorespiratory and muscular fitness; and psychosocial assessments (perceived physical activity barriers and social support).

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age; able to participate in aerobic and muscle-strengthening exercise; healthy (i.e., no diseases or clinical/mental health conditions which will prevent physical activity participation); does not meet minimum physical activity guidelines criteria for aerobic (≥ 150 minutes per week of moderate-to-vigorous intensity physical activity) and muscle-strengthening (≥ 2 days per week; 8-10 exercises for all major muscle groups) physical activity at time of enrollment; willing to be randomized to the intervention or control group.

Exclusion Criteria:

* less than 18 years old or greater than 35 years old; physical or mental health contradictions which do not allow participants to participate in physical activity; exceed minimum aerobic or muscle-strengthening physical activity guideline recommendations; unwilling to be randomized to either intervention or control group.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Change in objectively measured free-living physical activity | Baseline, 4 weeks (mid), and 8 weeks (end)
  7-day measurement using wrist-worn ActiGraph tri-axial accelerometer
Change in adherence to muscle-strengthening guidelines | Baseline, 4 weeks (mid), and 8 weeks (end)
  Assessed by 7-day physical activity recall interview to see if participants engaged in muscle-strengthening activity at least 2 days per week.

SECONDARY OUTCOMES:
Change in sleep quality | Baseline, 4 weeks (mid), and 8 weeks (end)
  7-day measurement using wrist-worn ActiGraph tri-axial accelerometer
Change in cardiorespiratory Fitness | Baseline, 4 weeks (mid), and 8 weeks (end)
  YMCA 3-minute step test
Change in muscular fitness | Baseline, 4 weeks (mid), and 8 weeks (end)
  60 second pushups and sit-ups muscular endurance tests (maximal repetitions)
Change in intrinsic Motivation | Baseline, 4 weeks (mid), and 8 weeks (end)
  Psychosocial survey
Change in social support | Baseline, 4 weeks (mid), and 8 weeks (end)
  Psychosocial survey
Change in perceived physical activity barriers | Baseline, 4 weeks (mid), and 8 weeks (end)
  Psychosocial survey
Change in body weight (kg) | Baseline, 4 weeks (mid), and 8 weeks (end)
  Measured using stadiometer to the nearest 0.1 kg
Height (cm | Baseline
  Measured using digital bodyweight scale to the nearest 0.1 cm
Change in body fat percentage | Baseline, 4 weeks (mid), and 8 weeks (end)
  Measured using the digital weight scale used to assess body weight via bioelectrical impedance

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J McDonough, M.S., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - Twin Cities, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDonough DJ, Helgeson MA, Liu W, Gao Z. Effects of a remote, YouTube-delivered exercise intervention on young adults' physical activity, sedentary behavior, and sleep during the COVID-19 pandemic: Randomized controlled trial. J Sport Health Sci. 2022 Mar;11(2):145-156. doi: 10.1016/j.jshs.2021.07.009. Epub 2021 Jul 24. PMID 34314877